CLINICAL TRIAL: NCT05123066
Title: Effect of Aquatic Training Versus Land Exercises on Motor Function in Children With Autism Spectrum Disorder
Brief Title: Effect of Aquatic Training on Motor Function in Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Mahmoud Abd-elmonem, Assist Prof. physical therapy for pediatric department, faculty of physical therappy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AQUATIC TRAINING
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2022-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Aquatic Therapy; Motor development; Land Exercises
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: They will be allocated randomly into two groups of equal numbers, group I (the aquatic training group) and the group II (land exercises).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquatic group (Experimental): group I
  Interventions: Other: Aquatic Exercises
- Land Exersises group (Experimental): group II
  Interventions: Other: Land Exercises

INTERVENTIONS:
Other: Aquatic Exercises — These 3 sets were the following:
  Set 1: warming up exercise as floating exercise 24 Set 2: Standing education/training Set 3: Walking education/training
  The exercises will be conducted taking in consideration safety measures as:
  1. Each participant will use Noodles to ensure safety.
  2. Each participant will train individually to ensure safety and avoid distraction.
  3. Each participant will use special swimming suit in case of lack of bowel and/or bladder control.
  Arms: Aquatic group
Other: Land Exercises — All participants were physical therapy intervention according to their level of functional impairment :
  Arms: Land Exersises group

SUMMARY:
Clinically, infants with Autism Spectrum Disorder often display gross motor delays in supine, prone, and sitting skills in their first year of life . Studies reveal that motor abnormalities in Autism Spectrum Disorder can occur very early in developmental trajectory.

DETAILED DESCRIPTION:
Hydrotherapy is an environment that may be conducive to encouraging physical activity in children with Autism Spectrum Disorder. The buoyancy of water can assist with movement, balance, and coordination .Water also provides an opportunity for social interaction through aquatic games and activities.Based on the literature, Aquatic therapy appears to be particularly beneficial for children with Autism Spectrum Disorder who need strong sensory stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 3 to 5 years.
* Mild to moderate autistic features according to GARS (scores from 60 to 110).

Exclusion Criteria:

* Significant visual or auditory defects.
* History of cerebral palsy or psychiatric disorder (e.g attention deficit hyperactivity disorder).
* Open wound.
* Dermatological diseases

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Autism Index | Treatment for 3 monthes
  Gilliam autism rating scale:
  Items on the developmental subscale address behaviors and milestones in the first 36 months of life. Items on the first three behavioral subscales are rated on a four point like scale ranging from Never Observed (0) to Frequently Observed (3). After completing it, the examiner calculated the total raw scores then converted into scaled scores and percentile ranks according to the examiner's manual. Higher scaled scores on a subscale represent severe autistic behavior. Finally, the total scaled scores were calculated to measure the autism index according to the examiner's manual. The higher the autism index, the higher the probability the individual has autism and the more severe the autistic behavior
Motor Development | Treatment for 3 monthes
  The Peabody Developmental Motor Scales-Second Edition:
  The gross motor function domain will be assessed in the current study. The gross motor function domains contain four subtests. Reflexes, Stationary ,Locomotion and Object Manipulation .
  Grading and Scoring of the PDMS-2 The therapist will ask the child to do a specific item and observes how the child is doing the task. Items are scored as 2, 1 or 0.
  0 = child cannot or will not attempt an item or the attempt does not indicate that the specific skill is emerging
  1. = child's performance shows a clear resemblance to item mastery criteria but does not fully meet the criteria or there are signs of an emerging skill
  2. = child performs item according to the criteria specified for mastering the skill
Pediatric Quality of life Inventory Scale | Treatment for 3 monthes
  Pediatric Quality of life Inventory Scale:
  The Arabic version will be used to assess quality of life. It contains questions about child's physical, emotional, social, and school functioning in the past 7 days. Parents/ child self-administered the quality of life after introductory instructions from the administrator. On the quality of life Generic Core Scales, for ease of interpretability, items are 22 reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better Health-Related quality of Life. To reverse score, transform the 0-4 scale items to 0-100 as follows: 0-100, 1=75, 2= 50, 3= 25 and 4= 0. Finally, the Scale Score for each dimension and Total Scale Score were calculated

CONTACTS AND LOCATIONS:
Overall Officials: Amira M ABD-ELMONEM, PhD, Study Chair — Department of Physical Therapy for Pediatrics, Faculty of Physical Therapy, Cairo University; MAI E ABBASS, PhD, Study Director — Department of Physical Therapy for Pediatrics, Faculty of Physical Therapy, Cairo University; AMR A OTHMAN, PhD, Study Director — Pediatrics Department, Faculty of Medicine, Sohag University
Locations (1):
- Eman S Albadry, Giza, Giza Governorate, Egypt